CLINICAL TRIAL: NCT04212442
Title: Improving Aging in Place for Older Adults in Subsidized Housing
Brief Title: Improving Aging in Place in Subsidized Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of California, Berkeley (Other); HumanGood (Other); University of Maryland, Baltimore (Other); Diocesan Housing Services Corporation of the Diocese of Camden, Inc (Other); Fair Share Housing Development (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rebecca Brown, M.D. MPH, Faculty - Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 831642; K76AG057016 (NIH)
Record Dates: First submitted 2019-12-16; First posted 2019-12-27 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Physical Disability; Cognitive Impairment; Physical Activity
Keywords: aging in place; physical activity; cognitive impairment; dementia; affordable housing; subsidized housing; functional impairment; home health aides; activities of daily living
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Dementia

STUDY DESIGN:
Intervention Model Description: This is a pilot study testing the adapted Function Focused Care intervention. The study employs a wait-list control design and site randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Upon enrollment, participants receive the adapted telephone-based intervention, the Independent Living Program for Affordable Housing, for two consecutive months.
  Interventions: Behavioral: Independent Living Program for Affordable Housing.
- Wait-list Control (Experimental): Two months after study enrollment, participants receive the adapted telephone-based intervention, the Independent Living Program for Affordable Housing, for two consecutive months.
  Interventions: Behavioral: Independent Living Program for Affordable Housing.

INTERVENTIONS:
Behavioral: Independent Living Program for Affordable Housing. — Two-month program intended to increase physical activity and function, including the following 4 steps:
  1. Environmental and Policy Assessments: Nurse facilitator works with the affordable housing staff to identify and recommend feasible interventions to alter the environment, policy, and procedures to optimize resident function and physical activity.
  2. Education: Nurse educates residents and study partners in the principles of the Independent Living Program, using established materials and adult learning techniques.
  3. Establishing Resident Goals: The nurse completes Capability Assessment Forms and helps resident set goals to increase function and physical activity.
  4. The nurse helps to motivate and mentor residents and study partners to achieve and maintain their goals, using evidence-based approaches.

SUMMARY:
This pilot study will evaluate the feasibility and preliminary effectiveness of an adapted version of the Function Focused Care intervention, delivered by telephone, for improving aging in place for older adults living in subsidized housing. The study will include participants with and without mild cognitive impairment or mild dementia and will examine whether the study outcomes differ by cognitive status. Findings from this study will provide new information about how to optimize function and physical activity among older adults with and without cognitive impairment living in subsidized housing.

DETAILED DESCRIPTION:
Millions of older adults with low incomes live in federally-subsidized housing and are at disproportionate risk for nursing home admission. Effective approaches are needed to improve aging in place for this vulnerable population. The objective of this study is to pilot test the feasibility and preliminary effectiveness of a telephone-based intervention to improve aging in place for older adults living in subsidized housing. In the first phase of this study, the investigators used methods of implementation science to adapt an existing intervention, Function Focused Care for Assisted Living, to the unique setting of affordable housing. Function Focused Care is a philosophy of care in which assisted living staff members engage residents in functional and physical activity during all care interactions. Prior research supports the effectiveness of Function Focused Care for maintaining function and increasing physical activity among older adults in assisted living settings.

In the first phase of this study, the investigators interviewed subsidized housing stakeholders - including residents, staff members, and caregivers - to identify barriers, facilitators, and needed adaptations to Function Focused Care for Assisted Living. The investigators used the findings from these interviews to adapt the intervention. In this 2-month pilot study, the investigators will use a wait-list control design with site randomization to assess the feasibility and preliminary effectiveness of the adapted intervention. The investigators will recruit individuals with and without mild cognitive impairment or mild dementia and will examine whether the study outcomes differ by cognitive status. The findings from this study will provide new information about how to optimize function and physical activity among older adults with and without cognitive impairment living in subsidized housing.

ELIGIBILITY:
Inclusion Criteria, Residents:

* Lives in an included subsidized housing setting
* 62 years of age or older
* Speaks English or Spanish well or very well
* Able to provide informed consent OR able to provide assent and has a proxy who provides informed consent on his/her behalf
* Has difficulty or needs help in at least 1 ADL and/or IADL OR has mild cognitive impairment or mild dementia based on their Montreal Cognitive Assessment (MoCA) score
* Not enrolled in hospice

Inclusion Criteria, Study Partners:

* Speaks English or Spanish well or very well
* Able to provide informed consent
* Spends at least an hour per week with the resident

Inclusion Criteria, Staff Members:

* Speaks English or Spanish well or very well
* Able to provide informed consent

Exclusion Criteria, Residents:

* Younger than 62 years of age
* Does not speak English or Spanish
* Lacks decision making capacity and lacks a proxy to consent on his/her behalf
* Does not have functional impairment or cognitive impairment
* Has moderate to severe dementia based on his/her MoCA score
* Is enrolled in hospice

Exclusion Criteria, Study Partners:

* Does not speak English or Spanish
* Unable to provide informed consent
* Does not spend at least an hour per week with the resident

Exclusion Criteria, Staff Members:

* Does not speak English or Spanish
* Unable to provide informed consent

Min Age: 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Brown, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (13):
- United States (13):
  - Northgate 2, Camden, New Jersey
  - Haven House, Cape May, New Jersey
  - Victorian Towers, Cape May, New Jersey
  - Stonegate 1, Pennsauken, New Jersey
  - Stonegate 2, Pennsauken, New Jersey
  - Mantua Presbyterian Apartments, Philadelphia, Pennsylvania
  - Old City Presbyterian Apartments, Philadelphia, Pennsylvania
  - Casa Carmen Aponte, Philadelphia, Pennsylvania
  - Neumann Senior Housing, Philadelphia, Pennsylvania
  - St. Francis VIlla, Philadelphia, Pennsylvania
  - Paschall Senior Housing, Philadelphia, Pennsylvania
  - Greenway Presbyterian Apartments, Philadelphia, Pennsylvania
  - Jackson Place, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Will share data based on request and following the development of an IPD sharing plan with the IRB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of the 3 year study period for the full parent study
Access Criteria: Identification of the purpose for wanting the data

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Apartment building
Groups:
- Immediate Intervention: Upon enrollment, participants receive the adapted telephone-based intervention, the Independent Living Program for Affordable Housing, for two consecutive months.
  Independent Living Program for Affordable Housing.: Two-month program intended to increase physical activity and function, including the following 4 steps:
  1. Environmental and Policy Assessments: Nurse facilitator works with the affordable housing staff to identify and recommend feasible interventions to alter the environment, policy, and procedures to optimize resident function and physical activity.
  2. Education: Nurse educates residents and study partners in the principles of the Independent Living Program, using established materials and adult learning techniques.
  3. Establishing Resident Goals: The nurse completes Capability Assessment Forms and helps resident set goals to increase function and physical activity.
  4. The nurse helps to motivate and mentor residents and study partners to achieve and maintain their goals, using evidence-based approaches.
- Wait-list Control: Two months after study enrollment, participants receive the adapted telephone-based intervention, the Independent Living Program for Affordable Housing, for two consecutive months.
  Independent Living Program for Affordable Housing.: Two-month program intended to increase physical activity and function, including the following 4 steps:
  1. Environmental and Policy Assessments: Nurse facilitator works with the affordable housing staff to identify and recommend feasible interventions to alter the environment, policy, and procedures to optimize resident function and physical activity.
  2. Education: Nurse educates residents and study partners in the principles of the Independent Living Program, using established materials and adult learning techniques.
  3. Establishing Resident Goals: The nurse completes Capability Assessment Forms and helps resident set goals to increase function and physical activity.
  4. The nurse helps to motivate and mentor residents and study partners to achieve and maintain their goals, using evidence-based approaches.
Period: Overall Study
Arm/Group | Immediate Intervention | Wait-list Control
Started | 47; 8 Apartment building | 28; 7 Apartment building
Completed | 42; 8 Apartment building | 23; 7 Apartment building
Not Completed | 5; 0 Apartment building | 5; 0 Apartment building

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Wait-list Control | Total
Number analyzed (Participants) | 47 | 28 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.9) | 72.3 (7.0) | 72.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 18 | 60
  Male | 5 | 10 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 30 | 2 | 32
  Black, non-Hispanic | 13 | 11 | 24
  Hispanic/Latino | 4 | 13 | 17
  Other (individuals who self-identified as American Indian or Alaska Native, Asian, or other race) | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 28 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in Precipitating Events Project (PEP) Functional Status Scale From Baseline to 2 Months for Immediate Intervention Sites and Waitlist Control Sites
Description: Self-reported ability to perform 7 ADLs, 5 IADLs, and 3 mobility tasks (Range, 0-30; higher scores indicate more functional impairment)
Time Frame: Baseline, 2 months
Population: Please note that due to loss to follow-up for self-reported outcome measures, the overall number of participants analyzed is not consistent with numbers provided in the rows in the participant flow module.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
score on a scale | -1.3 (1.7) | 0.6 (2.6)

2. Primary Outcome: Change in Short Physical Performance Battery Score From Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites
Description: Objective measure of lower extremity functioning in older adults (Range, 0-12; higher scores indicate worse lower extremity functioning)
  The measure will be collected only if in-person contact is possible during the COVID-19 outbreak.
Time Frame: Baseline, 2 months
Population: Unable to collect data due to visitation restrictions in the setting of the COVID pandemic
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Average Step Counts From Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites
Description: Measured using Fitbit
Time Frame: Measured continuously from 0-2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 42 | 23
steps | 9,706 (17,546) | 3,880 (17,186)

4. Primary Outcome: Change in Time Spent in Differing Levels of Activity From Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites
Description: Measured using Fitbit (minutes spent in each of 4 levels of activity: sedentary; lightly active; fairly active; very active)
Time Frame: Measured continuously from 0-2 months
Population: Please note that all data are missing due to a lack of synced Fitbit data.
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change in Physical Activity Scale for the Elderly (PASE) Score From Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites
Description: Self-reported physical activity (Range, 0-793; higher scores indicate greater physical activity)
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
score on a scale | 4.52 (38.95) | 16.25 (46.00)

6. Primary Outcome: Feasibility of Study Recruitment, Measured as Percentage of Eligible Participants Recruited
Description: Assessed using participant responses to invitation to participate in the study (enrolled vs. refused)
Time Frame: 0-4 months
Population: The count exceeds the number analyzed because this is a measure of eligible participants recruited by aim. In the immediate intervention arm, 54 eligible individuals were invited to participate of whom 7 declined and 47 were enrolled; for the waitlist control arm, 33 eligible individuals were invited to participate of whom 5 declined and 28 were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 54 | 33
Participants | 47 | 28

7. Primary Outcome: Feasibility of Study Retention, Measured as Percentage of Participants Retained Over Study Follow-up
Description: Assessed as percentage of participants who remain enrolled in the study
Time Frame: 0-4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 47 | 28
Participants | 42 | 23

8. Primary Outcome: Acceptability Assessed Using a Survey Question
Description: Self-reported acceptability of the intervention (5-point Likert scale ranging from very unacceptable (1) to very acceptable (5); higher numbers indicate higher acceptability)
Time Frame: 2 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
score on a scale | 4.0 [3.0 to 5.0] | 5.0 [4.0 to 5.0]

9. Primary Outcome: Number of Participants With High Fidelity to Treatment Protocol, Measured Using Fidelity Checklist
Description: Number of participants with >80% fidelity to treatment protocol, measured using fidelity checklist including each study protocol task
Time Frame: 0-4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 47 | 28
Participants | 37 | 21

10. Primary Outcome: Fidelity to Motivational Interviewing, Measured Using the Motivational Interviewing Treatment Integrity Scale (MITI 4)
Description: Assessed by psychologist (4 global scores, scored on a 5-point Likert scale from 1 (low) to 5 (high))
Time Frame: 2 months
Population: Please note that MITI scores were calculated at the level of the nurse providing motivational interviewing rather than at the level of the resident. Thus, only a single score is available for each group.
Measure: Median (Inter-Quartile Range); unit: 4 scores for subdomains
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 8 | 8
4 scores for subdomains
  Cultivating change | 4.0 [3.1 to 4.9] | 4.0 [3.1 to 4.9]
  Softening sustain | 3.8 [3.5 to 4.4] | 3.8 [3.5 to 4.4]
  Partnership | 4.3 [3.6 to 4.9] | 4.3 [3.6 to 4.9]
  Empathy | 4.3 [3.6 to 4.9] | 4.3 [3.6 to 4.9]

11. Secondary Outcome: Change in EuroQol 5 Dimensions (EQ-5D-5L) Scale From Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites
Description: Self-reported measure (Range, 11111-55555, converted to a single index utility score ranging from of 0-1; higher scores indicate better quality of life)
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
units on a scale | 0.09 (0.27) | -0.05 (0.34)

12. Secondary Outcome: Change in Geriatric Depression Scale Short Form (GDS Short Form) Score From Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites
Description: Self-reported measure of depressive symptoms (Range, 0-15; score of 5-8 suggests mild depression, 9-11 moderate depression, and 12-15 severe depression)
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 47 | 28
score on a scale | -1.26 (2.23) | 0.42 (2.02)

13. Secondary Outcome: Percentage of Participants With a Hospitalization During the Study Period (Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites)
Description: Self-reported hospitalization
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
Participants
  Baseline | 4 | 2
  Follow-up | 1 | 1

14. Secondary Outcome: Change in Number of Hospitalizations During the Study Period (Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites)
Description: Self-reported number of hospitalizations
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of hospitalizations
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
number of hospitalizations | -0.18 (0.61) | -0.08 (0.28)

15. Secondary Outcome: Percentage of Participants With an Emergency Department Visit During the Study Period (Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites)
Description: Self-reported emergency department visit
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
Participants
  Baseline | 5 | 6
  Follow-up | 7 | 3

16. Secondary Outcome: Change in Number of Emergency Department Visits During the Study Period (Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites)
Description: Self-reported number of emergency department visits
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
number of visits | 0.11 (0.74) | -0.38 (0.65)

17. Secondary Outcome: Percentage of Participants With a Move to a Higher Level of Care (Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites)
Description: Self-reported or emergency contact-reported move to a higher level of care, defined as a move to assisted living, board and care, or nursing home
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
Participants
  Baseline | 0 | 0
  Follow-up | 0 | 0

18. Secondary Outcome: Percentage of Participants With a Skilled Nursing Facility Stay (Baseline to 2 Months for Immediate Intervention and Waitlist Control Sites)
Description: Self-reported skilled nursing facility stay
Time Frame: Baseline, 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Wait-list Control
Number analyzed (Participants) | 28 | 13
Participants
  Baseline | 1 | 0
  Follow-up | 0 | 0

ADVERSE EVENTS:
Time Frame: 0-2 months
Arm/Group | Immediate Intervention | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/28
Other Adverse Events (participants affected / at risk) | 0/47 | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Intervention (N=47) | Wait-list Control (N=28)
Fall related to participating in intervention (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was conducted during the COVID pandemic. Due to challenges with participant follow-up in the setting of the pandemic, outcome data is missing for multiple participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04212442/Prot_SAP_000.pdf